CLINICAL TRIAL: NCT01102348
Title: Enhanced Protein-Energy Provision Via the Enteral Route in Critically Ill Patients: A Single Center Feasibility Trial of The PEP uP Protocol
Brief Title: Enhanced Protein-Energy Provision Via the Enteral Route in Critically Ill Patients
Acronym: PEP-uP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daren K. Heyland (Other)
Collaborators: Queen's University (Other); Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor-Investigator, Daren K. Heyland, Director of Clinical Evaluation Research Unit, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: PEP-uP Pilot
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Critically Ill
Keywords: Critically Ill; Nutrition Therapy; Enteral Nutrition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Before and after
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEP-uP Protocol (after) (Experimental): PEP-uP protocol and treatment algorithm implemented for all patients in ICU.
  Interventions: Other: PEP-uP Protocol
- Standard feeding protocol (before) (No Intervention): Enteral feeds are guided by a standard feeding protocol specified by pre-printed ICU admission orders. The admitting physician has the option of initiating the enteral feeding protocol or keeping the patient nil per os (NPO).

INTERVENTIONS:
Other: PEP-uP Protocol — Protocol documents (i.e. pre-printed order, algorithm for advancing feed, and algorithm for calculating rate of administering feed as per 24hour volume) and a slide presentation coupled with educational reminders (posters and bedside notices) and practice helps (tool to remind nurse to measure and report nutritional adequacy) were made available to all nurses, in bedside manuals and on the local intranet
  Arms: PEP-uP Protocol (after)

SUMMARY:
The purpose of this pilot study is to assess the feasibility, acceptability, and safety of a new feeding protocol, "The Enhanced Protein-Energy Provision via the Enteral Route in Critically Ill Patients: The PEP uP protocol."

DETAILED DESCRIPTION:
There is a well known and well described relationship between malnutrition, immune dysfunction, and infection. Critically ill patients are often hypermetabolic and can rapidly become nutritionally compromised. Repeated efforts over the past few years have not significantly improved the amount of calories delivered via the enteral route. Historically, feeding protocols have been used to guide the delivery of enteral nutrition (EN) but they frequently utilize conservative, reactionary approaches to optimizing nutrition.

We propose a new approach that protocolizes an aggressive approach to providing EN and shifts the paradigm from reactionary to proactive followed by de-escalation if nutrition therapy is not needed. The key components of this new protocol are the following: 1) Starting feeds at the target rate based on increasing evidence that some patients tolerate starting nutrition at higher rate of delivery and that slow start ups are not necessary. For patients who are hemodynamically stable, we propose to shift from an hourly rate target goal to a 24 hour volume goal and give nurses guidance on how to make up this volume if there was an interruption for non-gastrointestinal reasons. This 'volume-based' goal represents a significant shift in practice from traditional hourly rate goals in which nurses can increase the hourly rate depending on how many hours they have left in the day to ensure that the patient receives the 24 hour volume within the day. 2) For patients who are deemed unsuitable for high volume intragastric feeds, we provide an option to initiate 'trophic feeds' at a low volume of a concentrated feeding solution. By 'trophic', we mean a minimal volume of EN designed to maintain gastrointestinal structure and function, not designed to meet the patients caloric or protein needs. When deemed suitable, trophic feeds can be advanced to full feeds. 3) Rather than wait for a protein debt to accumulate because of inadequate delivery of EN, protein supplements are prescribed at initiation of EN and can be discontinued if EN is well tolerated. 4) We propose to start motility agents at the same time EN is started with a re-evaluation in the days following to see if it is necessary and we raised our gastric residual volume threshold from 200 to 250 ml. It has been shown in one randomized trial that a feeding protocol that starts a motility agent empirically at the time of initiation of feeds and uses a higher threshold for a critical gastric residual volume (250 ml) improves nutritional adequacy.

Since the bedside nurses initiate and utilize feeding protocols to achieve target goals, we will couple this newer generational feeding protocol with a comprehensive nurse-directed nutritional educational intervention that will focus on its safe and effective implementation. This focus on nursing nutrition education represents a major shift away from traditional education which has focused on dietitians and physicians.

We hypothesize that the combination of these components will safely improve the provision of energy and protein compared to usual care. We postulate that this increased provision of calories and protein may translate into improved clinical outcomes, particularly for the patients at the extremes of weight, but the current study is not powered to demonstrate such a difference. The purpose of this pilot study is to assess the feasibility, acceptability, and safety of this new feeding protocol, "The Enhanced Protein-Energy Provision via the Enteral Route in Critically Ill Patients: The PEP uP protocol."

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated within 48 hours of admission to the intensive care unit

Exclusion Criteria:

* Less than 72 hours in intensive care unit before discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of the feeding protocol | 10-12 months
  The primary outcome of this pilot study was the feasibility of the new feeding protocol as judged by a nursing questionnaire that evaluates their opinion of its safety and acceptability.

SECONDARY OUTCOMES:
Adequacy of EN | 10-12 months
  Calculated as proportion of EN received versus EN prescribed
Episodes of vomiting | 10-12 months
  Safety endpoints
Timeliness of initiation of EN | 10-12 months
  Actual timing of EN start
Episodes of aspiration | 10-12 months
  Safety end points
Episodes of aspiration & pneumonia | 10-12 months
  Safety end points

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, Principal Investigator — Clinical Evaluation Research Unit
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Heyland DK, Cahill NE, Dhaliwal R, Wang M, Day AG, Alenzi A, Aris F, Muscedere J, Drover JW, McClave SA. Enhanced protein-energy provision via the enteral route in critically ill patients: a single center feasibility trial of the PEP uP protocol. Crit Care. 2010;14(2):R78. doi: 10.1186/cc8991. Epub 2010 Apr 29. PMID 20429886